CLINICAL TRIAL: NCT03216954
Title: A Human Laboratory Study of n-Acetylcysteine for Alcohol Use Disorder
Brief Title: Influence of n-Acetylcysteine Maintenance on Alcohol Effects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: William Stoops (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, William Stoops, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BED IN 34; R21AA026129 (NIH)
Record Dates: First submitted 2017-07-07; First posted 2017-07-13 (Actual); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Subjects will receive oral placebo capsules two times daily.
  Interventions: Drug: Alcohol; Drug: Placebos
- Low Dose n-Acetylcysteine (Experimental): Subjects will receive 0.6 g oral n-acetylcysteine two times daily.
  Interventions: Drug: Alcohol; Drug: N-acetyl cysteine
- High Dose n-Acetylcysteine (Experimental): Subjects will receive 1.2 g oral n-acetylcysteine two times daily.
  Interventions: Drug: Alcohol; Drug: N-acetyl cysteine

INTERVENTIONS:
Drug: Alcohol — During each arm, subjects will receive doses of alcohol, designed to raise BALs to 0.015 and 0.03 g/dl.
Drug: Placebos — Subjects will receive placebo capsules
  Arms: Placebo
Drug: N-acetyl cysteine — Subjects will receive n-acetyl cysteine capsules
  Arms: High Dose n-Acetylcysteine; Low Dose n-Acetylcysteine

SUMMARY:
This study will evaluate the behavioral effects of alcohol during placebo and n-acetylcysteine maintenance using sophisticated human laboratory methods.

ELIGIBILITY:
Inclusion Criteria:

* able to speak/read English
* not seeking treatment at the time of the study
* one binge drinking episode (5+/4+ standard alcoholic drinks per drinking session for men and women, respectively) in the past 30 days
* recent alcohol use verified by ethyl glucuronide positive urine, as well as fulfillment of DSM-5 diagnostic criteria for alcohol use disorder
* ECG within normal limits
* otherwise healthy
* body mass index of 19-35
* females using an effective form of birth control and not pregnant or breast feeding
* judged by the medical staff to be psychiatrically and physically healthy
* able to abstain from alcohol for 12 hours prior to session
* no contraindications/allergies to n-acetylcysteine

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W Stoops, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then 1.2 g n-Acetylcysteine Then 2.4 g n-Acetylcysteine: Subjects were maintained on placebo for 5 days, then they were maintained on 1.2 g n-acetylcysteine daily for 5 days, then they were maintained on 2.4 g n-acetylcysteine for 5 days.
- 2.4 g n-Acetylcysteine Then 1.2 g n-Acetylcysteine Then Placebo: Subjects were maintained on 2.4 g n-acetylcysteine for 5 days, then they were maintained on 1.2 g n-acetylcysteine daily for 5 days, then they were maintained on placebo for 5 days.
- Placebo Then 2.4 g n-Acetylcysteine Then 1.2 g n-Acetylcysteine: Subjects were maintained on placebo for 5 days, then they were maintained on 2.4 g n-acetylcysteine, then they were maintained on 1.2 g n-acetylcysteine.
- 1.2 g n-Acetylcysteine Then Placebo Then 2.4 g n-Acetylcysteine: Subjects were maintained on 1.2 g n-acetylcysteine for 5 days, then they were maintained on placebo for 5 days, then they were maintained on 2.4 g n-acetylcysteine for 5 days.
- 1.2 g n-Acetylcysteine Then 2.4 g n-Acetylcysteine Then Placebo: Subjects were maintained on 1.2 g n-acetylcysteine for 5 days then they were maintained on 2.4 g n-acetylcysteine for 5 days, then they were maintained on placebo.
Period: Overall Study
Arm/Group | Placebo Then 1.2 g n-Acetylcysteine Then 2.4 g n-Acetylcysteine | 2.4 g n-Acetylcysteine Then 1.2 g n-Acetylcysteine Then Placebo | Placebo Then 2.4 g n-Acetylcysteine Then 1.2 g n-Acetylcysteine | 1.2 g n-Acetylcysteine Then Placebo Then 2.4 g n-Acetylcysteine | 1.2 g n-Acetylcysteine Then 2.4 g n-Acetylcysteine Then Placebo
Started | 4 | 3 | 3 | 3 | 1
Completed | 2 | 2 | 2 | 3 | 0
Not Completed | 2 | 1 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0
Not completed — Subject used cocaine during participation, which is an exclusion criterion. | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Completing subjects.
Groups:
- Crossover Study Drug Conditions: Subjects received oral placebo, 0.6 g n-acetylcysteine or 1.2 g n-acetylcysteine capsules two times daily. Dose condition was assigned in random order and all completing subjects received all dose conditions.
  Alcohol: During each condition, subjects received doses of alcohol, designed to raise BALs to 0.015 and 0.03 g/dl.
  Placebos: Subjects received placebo capsules. n-Acetylcysteine: Subjects received n-acetylcysteine capsules.
Arm/Group | Crossover Study Drug Conditions
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Alcohol Drinks Chosen
Description: The reinforcing effects of alcohol were determined using a self-administration procedure in which subjects choose to take previously sampled doses. Reinforcing effects are measured during maintenance on placebo and n-acetylcysteine.
Time Frame: After at least four days of placebo or n-acetylcysteine maintenance
Population: Completing Subjects
Measure: Mean (Standard Deviation); unit: Number of Alcohol Drinks Chosen
Groups:
- Placebo: Subjects received oral placebo capsules two times daily.
  Alcohol: During each arm, subjects will receive doses of alcohol, designed to raise BALs to 0.015 and 0.03 g/dl.
  Placebos: Subjects will receive placebo capsules
- Low Dose n-Acetylcysteine: Subjects received 0.6 g oral n-acetylcysteine two times daily.
  Alcohol: During each arm, subjects will receive doses of alcohol, designed to raise BALs to 0.015 and 0.03 g/dl.
  N-acetyl cysteine: Subjects will receive n-acetyl cysteine capsules
- High Dose n-Acetylcysteine: Subjects received 1.2 g oral n-acetylcysteine two times daily.
  Alcohol: During each arm, subjects will receive doses of alcohol, designed to raise BALs to 0.015 and 0.03 g/dl.
  N-acetyl cysteine: Subjects will receive n-acetyl cysteine capsules
Arm/Group | Placebo | Low Dose n-Acetylcysteine | High Dose n-Acetylcysteine
Number analyzed (Participants) | 9 | 9 | 9
Number of Alcohol Drinks Chosen | 3.1 (3.5) | 2.8 (3.5) | 3.8 (3.6)

ADVERSE EVENTS:
Time Frame: Full duration of each subject's participation, approximately 5 weeks.
Groups:
- Placebo Maintenance: Subjects received oral placebo capsules two times daily.
  Alcohol: During each arm, subjects will receive doses of alcohol, designed to raise BALs to 0.015 and 0.03 g/dl.
  Placebos: Subjects received placebo capsules
- 1.2 g n-Acetylcysteine Maintenance: Subjects received 0.6 g n-acetylcysteine capsules two times daily.
  Alcohol: During each arm, subjects will receive doses of alcohol, designed to raise BALs to 0.015 and 0.03 g/dl.
  Placebos: Subjects received placebo capsules n-Acetylcysteine: Subjects received 0.6 g n-acetylcysteine capsules
- 2.4 g n-Acetylcysteine Maintenance: Subjects received 1.2 g n-acetylcysteine capsules two times daily.
  Alcohol: During each arm, subjects will receive doses of alcohol, designed to raise BALs to 0.015 and 0.03 g/dl.
  Placebos: Subjects received placebo capsules n-Acetylcysteine: Subjects received 1.2 g n-acetylcysteine capsules
Arm/Group | Placebo Maintenance | 1.2 g n-Acetylcysteine Maintenance | 2.4 g n-Acetylcysteine Maintenance
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 1/14 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Maintenance (N=14) | 1.2 g n-Acetylcysteine Maintenance (N=14) | 2.4 g n-Acetylcysteine Maintenance (N=14)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — During placebo maintenance
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — During placebo maintenance
Blurry vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — during 1.2 g n-acetylcysteine/day maintenance
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — during 1.2 g n-acetylcysteine/day maintenance
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) — during 1.2 g n-acetylcysteine/day maintenance

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT03216954/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03216954/Prot_SAP_002.pdf